CLINICAL TRIAL: NCT01479868
Title: A Phase III Open-Label Study to Evaluate the Safety, Tolerability and Efficacy of TMC435 Plus PegIFNα-2a (Pegasys) and Ribavirin (Copegus) Triple Therapy in Chronic Hepatitis C Genotype-1 Infected Subjects Who Are Co-infected With Human Immunodeficiency Virus Type 1 (HIV-1)
Brief Title: A Study to Assess the Safety, Tolerability and Efficacy of TMC435 Along With Pegylated Interferon Alpha-2a (Pegasys) and Ribavirin (Copegus) Triple Therapy in Chronic Hepatitis C Genotype-1 Infected Patients Co-infected With Human Immunodeficiency Virus-Type 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR018334; TMC435-TiDP16-C212 (Other: Janssen Research & Development, LLC); NCT01727323 (obsolete NCT alias)
Record Dates: First submitted 2011-10-18; First posted 2011-11-28 (Estimated); Results first posted 2014-10-29 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Hepatitis C Virus Genotype-1
Keywords: Hepatitis C virus genotype-1; Human immunodeficiency virus-type 1; HCV-1; HIV-1; TMC435; Pegylated interferon alpha-2a; PegIFNα-2a; Pegasys; Ribavirin; RBV; Copegus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Simeprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TMC435 + pegylated interferon alpha-2a + ribavirin (Experimental): Patients will be administered TMC435 150 mg along with pegylated interferon alpha-2a 180 microgram and ribavirin 1000 or 1200 mg for 12 weeks. Pegylated interferon alpha-2a and ribavirin will only be continued until 24 to 48 weeks.
  Interventions: Drug: TMC435; Drug: Pegylated interferon alpha-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: TMC435 — TMC435 150 mg will be administered once daily for 12 weeks along with peginterferon alpha-2a and ribavirin.
Drug: Pegylated interferon alpha-2a — Pegylated interferon alpha-2a 180 microgram will be administered as subcutaneous injection of 0.5 mL until 24 to 48 weeks.
Drug: Ribavirin — Ribavirin 1000 or 1200 mg twice daily will be administered each day until 24 to 48 weeks.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of TMC435 along with pegylated interferon alpha-2a (PegIFNα-2a) and ribavirin (RBV) triple therapy in hepatitis C virus genotype-1 infected subjects, co-infected with human immunodeficiency virus-type 1, and to evaluate the number of patients with sustained virologic response (SVR) at 12 weeks after the planned end of treatment.

DETAILED DESCRIPTION:
This is an open-label (all the people know the identity of the intervention), single arm (study will be conducted in a single group) clinical study, to evaluate the safety, tolerability and efficacy of TMC435 along with pegylated interferon alpha-2a (PegIFNα-2a) and ribavirin (RBV) triple therapy in adult chronic hepatitis C (CHC) genotype-1 infected patients who are co-infected with human immunodeficiency virus-type 1 (HIV-1). The study consists of 3 phases, screening phase (Week -6), treatment phase, and a follow-up phase (up to 24 weeks). In the treatment phase, patients will be classified based on their experience with previous hepatitis C virus (HCV) treatment as follows: 1) HCV treatment-naive (patients who never received medication for the treatment of HCV); 2) prior HCV relapsers (patients who received at least 24 weeks of a PegIFNα-2a and RBV-based therapy and relapsed within 1 year after the last medication intake); and 3) prior HCV non-responders (can be further classified as, null responders: patients having at least 1 prior documented course of PegIFNα-2a and RBV therapy for at least 12 consecutive weeks; or partial responders: patients having at least 20 consecutive weeks which has not been discontinued due to intolerability to PegIFNα-2a and RBV therapy). All patients will receive TMC435 once daily along with PegIFNα-2a and RBV for 12 weeks. Patients who are continuing treatment only with PegIFNα-2a and RBV will follow until 24 or 48 weeks. Pharmacokinetics will be measured after collection of blood samples. Safety evaluations for adverse events, clinical laboratory tests, electrocardiogram, vital signs, physical examinations, and specific toxicities will be performed throughout the study. The total duration of treatment is approximately of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A liver biopsy required within 3 years prior to screening unless the patient has a contraindication for a liver biopsy
* Patients with bridging fibrosis or cirrhosis and without a liver biopsy result within 2 years prior screening must have an ultrasound taken within 2 months prior to the screening visit or during screening with no findings suspicious for hepatocellular carcinoma (HCC)
* Genotype-1 hepatitis C virus (HCV) infection
* Plasma HCV ribonucleic acid (RNA) of more than 10,000 IU per mL
* Documented human immunodeficiency virus-type 1 (HIV-1) infection at least 6 months prior to screening

Exclusion Criteria:

* Patient showing evidence of hepatic decompensation (ie, history or current evidence of ascites, bleeding varices or hepatic encephalopathy, albumin serum concentration less than 3.3 gm per dL, prolonged prothrombin time [PT] expressed as international normalized ratio [INR] more than 1.5)
* Any liver disease of non-HCV etiology
* Co-infection with hepatitis B virus (hepatitis B surface antigen [HBsAg] positive)
* An acute HIV-1 infection; or HIV-2 infection
* Change in antiretroviral (ARV) regimen within the last 4 weeks prior screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2011-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (32):
- United States (10):
  - Los Angeles, California
  - Washington D.C., District of Columbia
  - Orlando, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Newark, New Jersey
  - Albany, New York
  - New York, New York
  - Dallas, Texas
  - Houston, Texas
- Canada (2):
  - Toronto, Ontario
  - Montreal, Quebec
- France (4):
  - Lyon
  - Montpellier
  - Nantes
  - Paris
- Germany (7):
  - Berlin
  - Bonn
  - Cologne
  - Düsseldorf
  - Frankfurt
  - Freiburg im Breisgau
  - Hamburg
- Portugal (3):
  - Amadora
  - Lisbon
  - Porto
- San Juan, Puerto Rico
- Spain (3):
  - Badalona
  - Elche
  - Madrid
- United Kingdom (2):
  - Brighton
  - London

REFERENCES:
- [Derived] Andersohn F, Claes AK, Kulp W, Mahlich J, Rockstroh JK. Simeprevir with pegylated interferon alfa 2a plus ribavirin for treatment of hepatitis C virus genotype 1 in patients with HIV: a meta-analysis and historical comparison. BMC Infect Dis. 2016 Jan 11;16:10. doi: 10.1186/s12879-015-1311-3. PMID 26753774
- [Derived] Saeed S, Strumpf EC, Walmsley SL, Rollet-Kurhajec K, Pick N, Martel-Laferriere V, Hull M, Gill MJ, Cox J, Cooper C, Klein MB; Canadian Co-Infection Cohort Study; Cohen J, Conway B, Cooper C, Cote P, Cox J, Gill J, Haider S, Harris M, Haase D, Hull M, Montaner J, Moodie E, Pick N, Rachlis A, Rouleau D, Sandre R, Tyndall JM, Vachon ML, Walmsley S, Wong D. How Generalizable Are the Results From Trials of Direct Antiviral Agents to People Coinfected With HIV/HCV in the Real World? Clin Infect Dis. 2016 Apr 1;62(7):919-926. doi: 10.1093/cid/civ1222. Epub 2016 Jan 6. PMID 26743093
- [Derived] Dieterich D, Rockstroh JK, Orkin C, Gutierrez F, Klein MB, Reynes J, Shukla U, Jenkins A, Lenz O, Ouwerkerk-Mahadevan S, Peeters M, De La Rosa G, Tambuyzer L, Jessner W. Simeprevir (TMC435) with pegylated interferon/ribavirin in patients coinfected with HCV genotype 1 and HIV-1: a phase 3 study. Clin Infect Dis. 2014 Dec 1;59(11):1579-87. doi: 10.1093/cid/ciu675. Epub 2014 Sep 5. PMID 25192745

RESULTS

PARTICIPANT FLOW:
Groups:
- TMC435 150mg 12Wks PR24/48: Participants received TMC435, 150 mg once daily plus peginterferon alfa-2a (PegIFN alfa-2a) and ribavirin (RBV) for 12 Weeks, followed by PegIFN alfa-2a (P) and RBV (R) until Week 24/48 (PR24/48). Treatment was to be stopped at Week 24 for HCV treatment-naïve and prior HCV relapsers who met the response guided therapy criteria, and who did not have cirrhosis. All prior HCV non-responders (null and partial), participants with cirrhosis, and HCV treatment-naïve and prior HCV relapsers who did not meet the response guided therapy criteria had a 48-week treatment period.
Period: Overall Study
Arm/Group | TMC435 150mg 12Wks PR24/48
Started | 106 (Restricted to subject who received at least one dose of treatment (TMC435/RBV/PegIFN).)
Completed | 97
Not Completed | 9
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 4
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Not completed — Sponsor's Decision | 1
Not completed — Initiation of new HCV Therapy | 1

BASELINE CHARACTERISTICS:
Population: Analysis population included all participants who received at least 1 dose of study drug.
Arm/Group | TMC435 150mg 12Wks PR24/48
Number analyzed (Participants) | 106
Age, Continuous [Median (Full Range); unit: years] | 48 [27 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 90

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response at Week 12 (SVR 12)
Description: The SVR 12 was defined as hepatitis C virus (HCV) ribonucleic acid (RNA) levels less than (<) 25 international unit per milliliter (IU/mL) undetectable at the actual end of treatment (EOT), and HCV RNA levels <25 IU/mL undetectable or HCV RNA levels <25 IU/mL detectable at 12 Weeks after end of treatment.
Time Frame: 12 weeks after end of treatment (Week 24 or 48)
Population: Intent to treat (ITT) population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48
Number analyzed (Participants) | 106
percentage of participants | 73.6 [65.1 to 82.1]

2. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at Week 24 (SVR 24)
Description: The SVR 24 was defined as hepatitis C virus (HCV) ribonucleic acid (RNA) levels less than (<) 25 international unit per milliliter (IU/mL) undetectable at the actual end of treatment (EOT), and HCV RNA levels <25 IU/mL undetectable or HCV RNA levels <25 IU/mL detectable at 24 weeks after end of treatment.
Time Frame: 24 weeks after end of treatment (Week 24 or 48)
Population: The ITT population included all perticipants who had at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48
Number analyzed (Participants) | 106
percentage of participants | 72.6 [64.0 to 81.3]

3. Secondary Outcome: Percentage of Participants With Hepatitis C Virus Ribonucleic Acid (HCV-RNA) Less Than (<) 25 International Units (IU/mL) Undetectable or Detectable/Undetectable
Description: Percentage of participants with HCV RNA less than (<) 25 IU/mL undetectable (undet.) or detectable (det.)/undetectable at specific time points were observed.
Time Frame: Week 4, 12, 24, 36, and 48
Population: ITT population included all participants who had at least 1 dose of study drug. Here, "N" (number of participants analyzed) is the number of participants analyzed for this outcome measure, "n" is the number of participants analyzed for this outcome measure at specific time points.
Measure: Number; unit: percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48
Number analyzed (Participants) | 105
percentage of participants
  Week 4: < 25 IU/mL HCV-RNA undet. (n=105) | 65.7 [56.5 to 74.9]
  Week 4:< 25 IU/mL HCV-RNA det./undet. (n=105) | 88.6 [82.4 to 94.8]
  Week 12:< 25 IU/mL HCV-RNA undet. (n=97) | 94.8 [90.4 to 99.3]
  Week 12:< 25 IU/mL HCV-RNA det./undet. (n=97) | 97.9 [95.1 to 97.9]
  Week 24:< 25 IU/mL HCV-RNA undet. (n=90) | 90.0 [83.7 to 96.3]
  Week 24:< 25 IU/mL HCV-RNA det./undet. (n=90) | 93.3 [88.1 to 98.6]
  Week 48:< 25 IU/mL HCV-RNA undet. (n=20) | 100 [100 to 100]
  Week 48:< 25 IU/mL HCV-RNA det./undet. (n=20) | 100 [100 to 100]

4. Secondary Outcome: Percentage of Participants With On-treatment Failure
Description: Participants were considered as an on-treatment failure if, at actual end of treatment (EOT), there was confirmed detectable HCV RNA levels.
Time Frame: Week 1 to 48
Population: The ITT population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48
Number analyzed (Participants) | 106
percentage of participants | 17

5. Secondary Outcome: Percentage of Participants With Viral Breakthrough
Description: Confirmed increase of more than 1 log10 IU per mL in HCV RNA level from the lowest level reached, or a confirmed HCV RNA level of more than 100 IU per mL in participants whose HCV RNA levels had previously been below the limit of quantification (less than 25 IU per mL detectable) or undetectable (less than 25 IU per mL undetectable), while on study therapy.
Time Frame: Week 1 to 48
Population: The ITT population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48
Number analyzed (Participants) | 105
percentage of participants | 11.4

6. Secondary Outcome: Percentage of Participants With Viral Relapse
Description: Participants were considered to have a viral relapse when, at actual end of treatment, HCV RNA levels were less than 25 IU per mL undetectable; and during the follow-up period, HCV RNA levels were more than or equal to 25 IU per mL.
Time Frame: Week 1 to 72
Population: The ITT population included all participants who received at least 1 dose of study drug. Here, "N" (number of participants analyzed) is the number of participants analyzed for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48
Number analyzed (Participants) | 87
percentage of participants | 10.3

7. Secondary Outcome: Percentage of Participants With Normalized Alanine Aminotransferase Levels
Description: Participants with normalized alanine aminotransferase levels observed whose alanine aminotransferase levels were out of range at Baseline.
Time Frame: Baseline up to Week 72
Population: The ITT population included all participants who received at least 1 dose of study drug. Here "N" signifies participants evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48
Number analyzed (Participants) | 65
percentage of participants | 81.5

8. Secondary Outcome: Percentage of Human Immunodeficiency Virus (HIV) Participants With Virologic Failure
Description: Participants had confirmed HIV virologic failure if HIV viral load values were greater than or equal to 50 or 200 copies/mL among those who previously had less than 50 copies/mL.
Time Frame: Baseline to Week 72.
Population: Participants who received potent anti-HIV treatment with a combination of more than 3 anti-antiretroviral therapies to reduce HIV RNA viral load to undetectable levels were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48
Number analyzed (Participants) | 93
percentage of participants
  Greater than or equal to 50 copies/mL | 5.4
  Greater than or equal to 200 copies/mL | 2.2

9. Secondary Outcome: Mean Change From Baseline in Log10 Plasma Human Immunodeficiency Virus (HIV) Viral Load
Time Frame: Baseline (Day 1), Week 2, 4, 8, 12, 16, 20, 24, 28, 36, 42, 48, 52, 60 and 72
Population: Participants who received potent anti-HIV treatment with a combination of more than 3 antiretroviral therapies to reduce HIV RNA viral load to undetectable levels were analyzed. Here "n" signifies participants evaluable for this measure at specified time point.
Measure: Mean (Standard Deviation); unit: copies per milliliter
Arm/Group | TMC435 150mg 12Wks PR24/48
Number analyzed (Participants) | 93
copies per milliliter
  Baseline (n=93) | 1.3726 (0.25796)
  Change at Week 2 (n=91) | -0.0724 (0.23857)
  Change at Week 4 (n=93) | -0.0704 (0.25817)
  Change at Week 8 (n=92) | -0.0442 (0.40974)
  Change at Week 12 (n=90) | -0.0655 (0.30510)
  Change at Week 16 (n=88) | -0.0829 (0.23986)
  Change at Week 20 (n=86) | -0.0847 (0.25111)
  Change at Week 24 (n=88) | -0.0689 (0.24785)
  Change at Week 28 (n=82) | -0.0564 (0.26319)
  Change at Week 36 (n=85) | 0.0004 (0.24395)
  Change at Week 42 (n=35) | -0.0623 (0.29365)
  Change at Week 48 (n=79) | -0.0041 (0.36177)
  Change at Week 52 (n=36) | 0.0011 (0.20767)
  Change at Week 60 (n=40) | -0.0184 (0.20940)
  Change at Week 72 (n=38) | -0.0265 (0.18323)
  Change at End of study (n=93) | 0.0099 (0.33435)

10. Secondary Outcome: Mean Change From Baseline in CD4+ Cell Count
Time Frame: Baseline (Day 1), Week 2, 4, 8, 12, 16, 20, 24, 28, 36, 42, 48, 52, 60 and 72
Population: Participants who received potent anti-HIV treatment with a combination of more than 3 antiretroviral therapies to reduce HIV RNA viral load to undetectable levels were analyzed. Here, "n" is the number of participants analyzed for this outcome measure at spcific time points.
Measure: Mean (Standard Deviation); unit: cell counts per microliter
Arm/Group | TMC435 150mg 12Wks PR24/48
Number analyzed (Participants) | 93
cell counts per microliter
  Baseline (n=93) | 640.3 (243.11)
  Change at Week 2 (n=89) | -95.0 (190.34)
  Change at Week 4 (n=91) | -171.5 (170.67)
  Change at Week 8 (n=92) | -244.2 (185.04)
  Change at Week 12 (n=91) | -271.7 (194.49)
  Change at Week 16 (n=88) | -275.5 (183.96)
  Change at Week 20 (n=84) | -283.5 (175.27)
  Change at Week 24 (n=89) | -288.8 (202.31)
  Change at Week 28 (n=82) | -252.3 (203.45)
  Change at Week 36 (n=83) | -198.7 (225.62)
  Change at Week 42 (n=33) | -336.8 (240.64)
  Change at Week 48 (n=77) | -166.6 (248.25)
  Change at Week 52 (n=35) | -202.7 (222.89)
  Change at Week 60 (n=40) | -90.6 (189.74)
  Change at Week 72 (n=38) | -62.9 (175.61)
  Change at End of Study (n=93) | -51.1 (178.20)

11. Secondary Outcome: Change From Baseline in CD4+ Cell Count in Percentage
Time Frame: Baseline (Day 1), Week 2, 4, 8, 12, 16, 20, 24, 28, 36, 42, 48, 52, 60 and 72
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage of lymphocyte
Arm/Group | TMC435 150mg 12Wks PR24/48
Number analyzed (Participants) | 93
percentage of lymphocyte
  Baseline (n=93) | 31.65 (8.390)
  Change at Week 2 (n=89) | 0.42 (6.490)
  Change at Week 4 (n=91) | 2.50 (5.943)
  Change at Week 8 (n=92) | 3.85 (5.930)
  Change at Week 12 (n=91) | 3.93 (6.264)
  Change at Week 16 (n=88) | 5.47 (6.301)
  Change at Week 20 (n=84) | 5.27 (6.961)
  Change at Week 24 (n=89) | 5.50 (7.029)
  Change at Week 28 (n=82) | 3.79 (6.759)
  Change at Week 36 (n=83) | 2.75 (6.492)
  Change at Week 42 (n=33) | 6.41 (6.213)
  Change at Week 48 (n=77) | 2.09 (7.356)
  Change at Week 52 (n=35) | 3.26 (6.838)
  Change at Week 60 (n=40) | 0.25 (5.296)
  Change at Week 72 (n=38) | 0.70 (4.406)
  Change at End of study (n=93) | 0.13 (6.169)

12. Secondary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between administration of study drug and up to Day 126 that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Week 1 to Week 72
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | TMC435 150mg 12Wks PR24/48
Number analyzed (Participants) | 106
participants
  TEAEs | 102
  TESAEs | 6

ADVERSE EVENTS:
Time Frame: Week 1 to Week 72
Arm/Group | TMC435 150mg 12Wks PR24/48
Serious Adverse Events (participants affected / at risk) | 11/106
Other Adverse Events (participants affected / at risk) | 103/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TMC435 150mg 12Wks PR24/48 (N=106)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Anal haemorrhage (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
General physical health deterioration (General disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Catheter site infection (Infections and infestations) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Aspartate aminotransferase increased (Investigations) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TMC435 150mg 12Wks PR24/48 (N=106)
Fatigue (General disorders) | 48
Influenza like illness (General disorders) | 25
Asthenia (General disorders) | 24
Pyrexia (General disorders) | 12
Chills (General disorders) | 9
Injection site reaction (General disorders) | 8
Pain (General disorders) | 7
Injection site erythema (General disorders) | 6
Insomnia (Psychiatric disorders) | 27
Mood altered (Psychiatric disorders) | 20
Depression (Psychiatric disorders) | 19
Anxiety (Psychiatric disorders) | 13
Sleep disorder (Psychiatric disorders) | 6
Nausea (Gastrointestinal disorders) | 31
Diarrhoea (Gastrointestinal disorders) | 25
Vomiting (Gastrointestinal disorders) | 14
Constipation (Gastrointestinal disorders) | 12
Neutropenia (Blood and lymphatic system disorders) | 33
Anaemia (Blood and lymphatic system disorders) | 30
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Headache (Nervous system disorders) | 35
Dizziness (Nervous system disorders) | 13
Pruritus (Skin and subcutaneous tissue disorders) | 19
Dry skin (Skin and subcutaneous tissue disorders) | 16
Eczema (Skin and subcutaneous tissue disorders) | 8
Alopecia (Skin and subcutaneous tissue disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 15
Back pain (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9
Decreased appetite (Metabolism and nutrition disorders) | 21
Weight decreased (Investigations) | 13
Neutrophil count decreased (Investigations) | 6
Nasopharyngitis (Infections and infestations) | 7
Upper respiratory tract infection (Infections and infestations) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less